CLINICAL TRIAL: NCT03028532
Title: Administration of Clomiphene: Short and Long Term Metabolism in an Anti-Doping Setting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stuart Willick (Other)
Collaborators: Sports Medicine Research and Testing Laboratory (Industry); Partnership for Clean Competition (Other)
Responsible Party: Sponsor-Investigator, Stuart Willick, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 97194
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Sports Drug Abuse; Abuse of Steroids or Hormones
Keywords: Healthy Volunteers; Sports Medicine; Anti-doping; Athletes; Men's Health
MeSH Terms: interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clomid (Experimental): All participants will be receiving Clomid and will follow the same study procedures.
  Interventions: Drug: Clomid

INTERVENTIONS:
Drug: Clomid — Participants will self-administer Clomid (50mg oral tablet) once daily for 30 consecutive days
  Other Names: Clomiphene; Clomifene

SUMMARY:
Clomiphene (Clomid) is a drug FDA approved to treat female infertility, however, it is often used by men in an off-label setting to both treat male infertility and in a multitude of sports disciplines to increase performance.

Study Objectives:

* Determine detection windows for clomiphene and its metabolites in urine following a medium-term administration
* Understand the effect of clomiphene administration on luteinizing hormone (LH), follicle-stimulating hormone (FSH), and serum testosterone (T) concentrations in a longitudinal manner
* Identify changes in current steroidal module of Athlete Biological Passport

DETAILED DESCRIPTION:
Clomiphene, pharmaceutically prepared as clomiphene citrate, is a selective estrogen receptor modulator (SERM) with a therapeutic indication to treat female infertility. Though FDA-approved only for use in women, clomiphene is often prescribed off-label to males to treat male infertility and secondary hypogonadism due to its ability to increase serum testosterone levels. Numerous clinical studies have documented both the effectiveness for these indications and safety of clomiphene administration in males. Increasing the concentration of circulating testosterone can have additional effects, including the enhancement of performance in sports. As such, clomiphene is already abused by athletes in several sporting disciplines, including mixed martial arts, cycling, and bodybuilding. Therefore, clomiphene is a prohibited substance under the World Anti-Doping Agency code . Though the parent compound and metabolites of clomiphene are directly detectable in routine anti-doping screening, the urinary detection window and the effect of clomiphene administration on other anti-doping markers are unknown and thus the foci of this study.

ELIGIBILITY:
Inclusion Criteria:

- Active males who engage in regular exercise between the ages of 18 and 40 on the day of enrollment

• For this study, regular exercise is defined as: physical activity resulting in an increased heart rate for at least 30 minutes per day, 4-5 days per week.

Exclusion Criteria:

* Individuals outside of the described age range on the day of enrollment
* Individuals who are in a Registered Testing Pool for anti-doping purposes, or individuals who for any reason could be subject to doping control testing
* Individuals who are unwilling or unable to provide blood or urine samples
* Individuals who do not actively exercise
* Individuals with any history of cancer, cardiovascular disease, endocrine abnormalities, infertility, hypoandrogenism, renal disease, hepatic disease, neurologic disease, or any psychiatric history
* Individuals who have previously used anabolic steroids, selective estrogen receptor modulators (SERMs), selective androgen receptor modulators (SARMs), or who are currently using any substances included on the WADA Prohibited List
* History of venous thromboembolic disease (i.e. deep vein thrombosis or pulmonary embolism)
* History of untreated cataracts
* History of intracranial lesions such as pituitary tumors
* Transaminase elevation greater than 3 times the upper limit of normal (ULN)
* Moderate or heavy alcohol intake

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
The window of detection for the clomiphene parent compound and metabolites following a 30-day administration will be identified. | Day 30 through end of study participation (minimum, Day 72)
  ◦This will be determined as the amount of time following the final dose (day 30) until clomiphene nor its metabolites are no longer detectable in a urine sample.

SECONDARY OUTCOMES:
Effect of clomiphene administration on serum LH, FSH, and T levels for potential inclusion into a hematological-based longitudinal steroid profile. | Day 30 through end of study participation (minimum, Day 72)
  A baseline for LH, FSH, and T will be established using the average of serum concentrations calculated from the pre-administration samples from each subject.The change in serum concentrations following administration will be compared against the baseline values.
Effect on current steroidal module of Athlete Biological Passport | Day 30 through end of study participation (minimum, Day 72)
  ◦The steroidal module of the Athlete Biological Passport, a statistical model used to identify doping, will be used for data analysis in this study.As stated in the ABP Operating Guidelines, the steroidal compounds described above are considered for the ABP steroidal module in addition to the following ratios: T/E, A/T, A/Etio, 5aAdiol/5βAdiol, and 5aAdiol/E. Changes in the urinary steroid concentrations and these ratios will be assessed over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Willick, MD, Principal Investigator — University of Utah
Locations (1):
- Heidi Jo Hansen, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guay AT, Jacobson J, Perez JB, Hodge MB, Velasquez E. Clomiphene increases free testosterone levels in men with both secondary hypogonadism and erectile dysfunction: who does and does not benefit? Int J Impot Res. 2003 Jun;15(3):156-65. doi: 10.1038/sj.ijir.3900981. PMID 12904801
- [Background] Katz DJ, Nabulsi O, Tal R, Mulhall JP. Outcomes of clomiphene citrate treatment in young hypogonadal men. BJU Int. 2012 Aug;110(4):573-8. doi: 10.1111/j.1464-410X.2011.10702.x. Epub 2011 Nov 1. PMID 22044663
- [Background] Niederberger C. Re: outcomes of clomiphene citrate treatment in young hypogonadal men. J Urol. 2013 Mar;189(3):1039. doi: 10.1016/j.juro.2012.11.143. Epub 2013 Jan 22. No abstract available. PMID 23394666
- [Background] Taylor F, Levine L. Clomiphene citrate and testosterone gel replacement therapy for male hypogonadism: efficacy and treatment cost. J Sex Med. 2010 Jan;7(1 Pt 1):269-76. doi: 10.1111/j.1743-6109.2009.01454.x. Epub 2009 Aug 17. PMID 19694928
- [Background] Chandrapal JC, Nielson S, Patel DP, Zhang C, Presson AP, Brant WO, Myers JB, Hotaling JM. Characterising the safety of clomiphene citrate in male patients through prostate-specific antigen, haematocrit, and testosterone levels. BJU Int. 2016 Dec;118(6):994-1000. doi: 10.1111/bju.13546. Epub 2016 Jun 24. PMID 27226135
- [Background] Helo S, Mahon J, Ellen J, Wiehle R, Fontenot G, Hsu K, Feustel P, Welliver C, McCullough A. Serum levels of enclomiphene and zuclomiphene in men with hypogonadism on long-term clomiphene citrate treatment. BJU Int. 2017 Jan;119(1):171-176. doi: 10.1111/bju.13625. Epub 2016 Sep 11. PMID 27511863
- [Background] Moskovic DJ, Katz DJ, Akhavan A, Park K, Mulhall JP. Clomiphene citrate is safe and effective for long-term management of hypogonadism. BJU Int. 2012 Nov;110(10):1524-8. doi: 10.1111/j.1464-410X.2012.10968.x. Epub 2012 Mar 28. PMID 22458540
- [Background] Patel DP, Brant WO, Myers JB, Presson AP, Johnstone EB, Dorais JA, Aston KI, Carrell DT, Hotaling JM. The safety and efficacy of clomiphene citrate in hypoandrogenic and subfertile men. Int J Impot Res. 2015 Nov-Dec;27(6):221-4. doi: 10.1038/ijir.2015.21. Epub 2015 Aug 20. PMID 26289907
- [Background] Roth LW, Ryan AR, Meacham RB. Clomiphene citrate in the management of male infertility. Semin Reprod Med. 2013 Jul;31(4):245-50. doi: 10.1055/s-0033-1345271. Epub 2013 Jun 17. PMID 23775379
- [Derived] Miller GD, Moore C, Nair V, Hill B, Willick SE, Rogol AD, Eichner D. Hypothalamic-Pituitary-Testicular Axis Effects and Urinary Detection Following Clomiphene Administration in Males. J Clin Endocrinol Metab. 2019 Mar 1;104(3):906-914. doi: 10.1210/jc.2018-01159. PMID 30295816
- See also: Clomid Drug Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2012/016131s026lbl.pdf
- See also: USADA Sanctions — http://www.usada.org/testing/results/sanctions/
- See also: Clomid Drug Information — http://www.evolutionary.org/clomid-clomiphene-citrate
- See also: Clomid Use in MMA — http://www.mmafighting.com/2016/7/23/12261944/brock-lesnar-tested-positive-for-anti-estrogen-lesnar-jon-jones-won-t